CLINICAL TRIAL: NCT05521620
Title: What Effect Does a Father-friendly NICU Have on Children, Parents, and Staff?
Brief Title: A Father-friendly Neonatal Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kolding Sygehus (Other)
Responsible Party: Principal Investigator, Betty Nørgaard, Principal Investigator, Kolding Sygehus
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 19/20297
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Stress; Self Efficacy; Perception, Self
Keywords: Father; Intensive Care Units, Neonatal; Parental support; Stress; Self-efficacy; Mothers; Nurse; Participatory reseach; Masculinity
MeSH Terms: conditions — Masculinity

STUDY DESIGN:
Intervention Model Description: A before- and-after intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Father-friendly NICU (Active Comparator): * Fathers have skin-to-skin contact with their infants
  * Fathers participate in important situations
  * Fathers receive information and guidance directly
  * Both parents participate in meaningful conversations
  * The department organize mother and father groups
  * The families have the opportunity to have a close family member to support them
  * Older siblings have the opportunity to stay overnight.
  * The department offer counseling by a social worker
  Interventions: Behavioral: The father-friendly NICU
- No Father-friendly NICU (baseline) (No Intervention): Baseline - before implementation of the intervention

INTERVENTIONS:
Behavioral: The father-friendly NICU — * Fathers have skin-to-skin contact with their infants
  * Fathers participate in important situations
  * Fathers receive information and guidance directly
  * Both parents participate in meaningful conversations
  * The department organize mother and father groups
  * The families have the opportunity to have a close family member to support them
  * Older siblings have the opportunity to stay overnight.
  * The department offer counseling by a social worker
  Arms: Father-friendly NICU

SUMMARY:
An early parent-child relationship is important for a child's development, both intellectually and socially. The admission of premature or ill newborns to neonatal intensive care units (NICUs) may make the establishment of the parent-child relationship challenging due to parents' anxiety and despair.

Traditionally, most healthcare professionals have mainly focused on infants and mothers, even though fathers often feel stressed, powerless, and helpless, and find it difficult to establish a father-child relationship. The aim of this study is to investigate the effect of a father-friendly NICU on infants, parents and staff.

DETAILED DESCRIPTION:
An early parent-child relationship is important for a child's development, both intellectually and socially. The admission of premature or ill newborns to neonatal intensive care units (NICUs) may make the establishment of the parent-child relationship challenging due to parents' anxiety and despair.

Traditionally, most healthcare professionals have mainly focused on infants and mothers, even though fathers often feel stressed, powerless, and helpless, and find it difficult to establish a father-child relationship. The aim of this study is to investigate the effect of a father-friendly NICU on infants, parents and staff.

The study was conducted in 3 steps

1. A baseline measurement
2. Development and implementation of the intervention a father friendly NICU
3. After measurement

Different questionnaires were used:

* The Parental Stressor Scale: Neonatal Intensive Care Unit (PSS:NICU)
* The Nurse Parent Support Tool (NPST)
* A questionnaire intended to measure nurses self-efficacy (SE).

The study was approved by the Danish Data Protection Agency (No 19/20297) and the procedures were in accordance with the Helsinki Declaration. In accordance with the Danish law, this study did not need to be reviewed by an ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* fathers/mothers with infants admitted to the NICU were eligible
* nurses who work in Danish NICUs

Exclusion Criteria:

* fathers/mothers who did not understand verbal and written Danish
* fathers/mothers of critically ill newborn infants
* fathers of newborn infants whose mother was critically ill
* fathers/mothers of newborn infants admitted to the NICU from home.
* nurses without patient-contact, on maternity- or long-term sickness-leave

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — mother and father
Enrollment: 500 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Stress (The Parental Stressor Scale: Neonatal Intensive Care Unit) | Measured on admission to the NICU (during the first 3 days of hospitalization), at the 14th day of hospitalization , and at the day of discharge from the NICU (up to 1/2 year)
  The primary outcome was the difference in the overall stress score, determined using the Parental Stressor Scale: Neonatal Intensive Care Unit (PSS:NICU) score in both the control and intervention groups.
  Fathers were asked to rate their stress related to particular situations on a 5-point Likert scale, ranging from 1 (not at all stressful) to 5 (extremely stressful). Fathers who had not experienced a particular situation on an item indicated this with a "not relevant" response. The maximal score was 5, a high score indicating a high level of paternal stress.
Parental Support (The Nurse Parent Support Tool) | Measured on admission to the NICU (during the first 3 days of hospitalization), and at the day of discharge from the NICU (up to 1/2 year)
  The primary outcome was the difference in fathers' perception of received staff support in the control group compared to the intervention group.
  The questionnaire included four dimensions of nurse support: 1) communication of information related to the infant's condition and care (nine items), 2) support mainly directed to enhance parental role (four items), 3) emotional support to help parents cope with their infant's sickness (three items), and 4) caregiving support concerning the quality of care provided to the infant (five items).
  For each item, the parents indicated the degree of support on a 5-point Likert scale ranging from 1 (never) to 5 (always) 19.
Nurses self-efficacy (Self-efficacy (SE)) | Before the start of the development of the intervention (August 2011) till 18 months after the implementation of the intervention (January 2015)
  The primary outcome was the difference between the nurses' SE scores for father and mother questions in the intervention group in comparison with the control group
  The nurses were asked to evaluate own ability to guide and support the parents in different situations (Self-efficacy score). The SE score was rated on a scale ranging from 1, indicating "Not at all sure," to 10, indicating "Definitely sure".
Self-efficacy follow-up | After the implementation of the intervention (January 2015) to five years after (February 2021).
  The primary outcome was the difference between the nurses' SE score on father and mother questions from after the implementation of the intervention to five years after.
  The nurses were asked to evaluate own ability to guide and support the parents in different situations (Self-efficacy score). The SE score was rated on a scale ranging from 1, indicating "Not at all sure," to 10, indicating "Definitely sure".

CONTACTS AND LOCATIONS:
Overall Officials: Betty Noergaard, Ph.d, Principal Investigator — Department of Paediatrics and Adolescent Medicine, Lillebaelt Hospital,Kolding
Locations (1):
- Department of Paediatrics and Adolescent Medicine at the University Hospital of Southern Denmark, Kolding, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: Yes
all individual patient data (IPD) that underlie results in a publication
Supporting Information: SAP
Time Frame: Ending 5 years following article publication.

REFERENCES:
- [Background] Meberg A, Wataker H. [Family-focused neonatal care]. Tidsskr Nor Laegeforen. 2010 Sep 9;130(17):1730-1. doi: 10.4045/tidsskr.10.0293. No abstract available. Norwegian. PMID 20835285
- [Background] Fegran L, Helseth S, Fagermoen MS. A comparison of mothers' and fathers' experiences of the attachment process in a neonatal intensive care unit. J Clin Nurs. 2008 Mar;17(6):810-6. doi: 10.1111/j.1365-2702.2007.02125.x. PMID 18279284
- [Background] Lindberg B, Axelsson K, Ohrling K. Adjusting to being a father to an infant born prematurely: experiences from Swedish fathers. Scand J Caring Sci. 2008 Mar;22(1):79-85. doi: 10.1111/j.1471-6712.2007.00563.x. PMID 18269426
- [Background] Sullivan JR. Development of father-infant attachment in fathers of preterm infants. Neonatal Netw. 1999 Oct;18(7):33-9. doi: 10.1891/0730-0832.18.7.33. PMID 10808886
- [Background] Mackley AB, Locke RG, Spear ML, Joseph R. Forgotten parent: NICU paternal emotional response. Adv Neonatal Care. 2010 Aug;10(4):200-3. doi: 10.1097/ANC.0b013e3181e946f0. PMID 20697219
- [Background] Pohlman S. Fathering premature infants and the technological imperative of the neonatal intensive care unit: an interpretive inquiry. ANS Adv Nurs Sci. 2009 Jul-Sep;32(3):E1-16. doi: 10.1097/ANS.0b013e3181b0d68c. PMID 19707083
- [Background] Lundqvist P, Westas LH, Hallstrom I. From distance toward proximity: fathers lived experience of caring for their preterm infants. J Pediatr Nurs. 2007 Dec;22(6):490-7. doi: 10.1016/j.pedn.2007.04.008. PMID 18036470
- [Background] Kaaresen PI, Ronning JA, Ulvund SE, Dahl LB. A randomized, controlled trial of the effectiveness of an early-intervention program in reducing parenting stress after preterm birth. Pediatrics. 2006 Jul;118(1):e9-19. doi: 10.1542/peds.2005-1491. PMID 16818541
- [Background] Pohlman S. The primacy of work and fathering preterm infants: findings from an interpretive phenomenological study. Adv Neonatal Care. 2005 Aug;5(4):204-16. doi: 10.1016/j.adnc.2005.03.002. PMID 16084478
- [Background] Franck LS, Spencer C. Parent visiting and participation in infant caregiving activities in a neonatal unit. Birth. 2003 Mar;30(1):31-5. doi: 10.1046/j.1523-536x.2003.00214.x. PMID 12581037
- [Background] Lundqvist P, Jakobsson L. Swedish men's experiences of becoming fathers to their preterm infants. Neonatal Netw. 2003 Nov-Dec;22(6):25-31. doi: 10.1891/0730-0832.22.6.25. PMID 14700179
- [Background] Miles MS, Holditch-Davis D. Parenting the prematurely born child: pathways of influence. Semin Perinatol. 1997 Jun;21(3):254-66. doi: 10.1016/s0146-0005(97)80067-5. PMID 9205979
- [Background] Ortenstrand A, Westrup B, Brostrom EB, Sarman I, Akerstrom S, Brune T, Lindberg L, Waldenstrom U. The Stockholm Neonatal Family Centered Care Study: effects on length of stay and infant morbidity. Pediatrics. 2010 Feb;125(2):e278-85. doi: 10.1542/peds.2009-1511. Epub 2010 Jan 25. PMID 20100748
- [Background] Johnson AN. Engaging fathers in the NICU: taking down the barriers to the baby. J Perinat Neonatal Nurs. 2008 Oct-Dec;22(4):302-6. doi: 10.1097/01.JPN.0000341361.37822.34. PMID 19011495
- [Background] Arockiasamy V, Holsti L, Albersheim S. Fathers' experiences in the neonatal intensive care unit: a search for control. Pediatrics. 2008 Feb;121(2):e215-22. doi: 10.1542/peds.2007-1005. Epub 2008 Jan 8. PMID 18182470
- [Background] Novak JC. Facilitating nurturant fathering behavior in the NICU. J Perinat Neonatal Nurs. 1990 Sep;4(2):68-77. doi: 10.1097/00005237-199009000-00009. PMID 2391649
- [Background] Levy-Shiff R, Hoffman MA, Mogilner S, Levinger S, Mogilner MB. Fathers' hospital visits to their preterm infants as a predictor of father-infant relationship and infant development. Pediatrics. 1990 Aug;86(2):289-93. PMID 2371105
- [Background] Bogdan R, Brown MA, Foster SB. Be honest but not cruel: staff/parent communication on a neonatal unit. Hum Organ. 1982 Spring;41(1):6-16. doi: 10.17730/humo.41.1.03x7x4214201v7p2. No abstract available. PMID 10254504
- [Background] Ammentorp J, Kofoed PE. Coach training can improve the self-efficacy of neonatal nurses. A pilot study. Patient Educ Couns. 2010 May;79(2):258-61. doi: 10.1016/j.pec.2009.08.015. Epub 2009 Sep 27. PMID 19786336
- [Background] Reid M, Lloyd D, Campbell G, Murray K, Porter M. Scottish neonatal intensive care units; a study of staff and parental attitudes. Health Bull (Edinb). 1995 Sep;53(5):314-25. PMID 7490204
- [Result] Noergaard B, Ammentorp J, Garne E, Fenger-Gron J, Kofoed PE. Fathers' Stress in a Neonatal Intensive Care Unit. Adv Neonatal Care. 2018 Oct;18(5):413-422. doi: 10.1097/ANC.0000000000000503. PMID 29746269
- [Result] Noergaard B, Ammentorp J, Fenger-Gron J, Kofoed PE, Johannessen H, Thibeau S. Fathers' Needs and Masculinity Dilemmas in a Neonatal Intensive Care Unit in Denmark. Adv Neonatal Care. 2017 Aug;17(4):E13-E22. doi: 10.1097/ANC.0000000000000395. PMID 28749826
- [Result] Noergaard B, Johannessen H, Fenger-Gron J, Kofoed PE, Ammentorp J. Participatory Action Research in the Field of Neonatal Intensive Care: Developing an Intervention to Meet the Fathers' Needs. A Case Study. J Public Health Res. 2016 Dec 21;5(3):744. doi: 10.4081/jphr.2016.744. eCollection 2016 Dec 9. PMID 28083521